CLINICAL TRIAL: NCT02504385
Title: The Effect of Timocco's Virtual Reality Environment on the Motor Functioning and Participation Abilities Among Children With DCD
Brief Title: The Effect of Virtual Reality on Motor Functioning and Participation Abilities Among Children With DCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Timocco Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COM 0024-14
Record Dates: First submitted 2015-03-29; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality Timocco (Experimental): The study group will integrate the use of Timocco in occupational therapy sessions. The session will begin with 15 minutes of spatial activity involving sensory-motor practice, 15 minutes of activity in a virtual environment, and 15 minutes of structured activity at a desk.
  Interventions: Device: Virtual Reality Timocco
- Conventional OT intervention (Active Comparator): The control group will be given conventional occupational therapy without using Timocco. In order to ensure that the therapy sessions in this group have a structure similar to that one used in the study group, each session will include 25 to 30 minutes of spatial sensory-motor activity, followed by 15 to 20 minutes of structured practice at a desk.
  Interventions: Other: Conventional OT intervention

INTERVENTIONS:
Device: Virtual Reality Timocco — Timocco virtual reality system is a motion based comuter games that was designed for child development therpay. The children will play Timocco for 15 minutes every session.
  Arms: Virtual Reality Timocco
Other: Conventional OT intervention — Traditional Occupational Therapy intervention will be givven to the control group.
  Arms: Conventional OT intervention

SUMMARY:
The subjet of this study is to explore the effect of using virtual reality environment at the clinic and at home (using Timocco) on the motor and participation abilities of children with DCD (Developmental Coordination Disorder).

The study will examine the efficacy of using virtual reality gaming environment (Timocco) for treating children with DCD and the use of remote therapy, by shifting the focus of therapy from the clinic to the home environment, using the remote control system of Timocco for home practice.

DETAILED DESCRIPTION:
The efficacy of using VR (Virtual Reality) as a therapeutic tool as an integral part of Occupational Therapy intervention will be examined in this study. The study will be conducted in two stages: the first will be conducted at the Child Development Center of the Clalit HMO (Health Maintenance Organization), and the second will take place in the child's home.

The first intervention will take approximately 8 to 10 weeks, during which eight data collection sessions will be conducted, each of 45 minutes duration.

The study group will integrate the use of Timocco in occupational therapy sessions while the control group will be given conventional occupational therapy without using Timocco.

In the second intervention, the study group will be given access to the virtual-reality environment of Timocco to be used at home, and will not include therapy sessions at the Child Development Center. An assessment before and after intervention will be held for both groups for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Children,
* native Hebrew speakers, between the ages of 4 and 6 diagnosed with DCD.

Exclusion Criteria:

* Children with complicated special needs (e.g., limited cognitive abilities, CP, ASD),
* children who received occupational or physical therapy interventions in the last 12 months.

Ages: 4 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The score in Motor and participation assessments (Henderson, S. & Sugden, D. 1992) | up to 18 weeks
Score in Timocco virtual reality system (number of wrong moves; Correct moves;response time) | up to 18 weeks
  data will be gathered using Timocco for the entire intervention

SECONDARY OUTCOMES:
DCD-Q (BN. Wilson, BJ. Kaplan, SG. Crawford and G. Roberts, 2009) | up to 18 weeks
  The questionnaire will be filled once at the beginning, once again at the end of phase 1 (in the clinic) , and last time after home practice (the second phase).
Participation questionnaire (Yarus, 2010) | up to 18 weeks
  The questionnaire will be filled once at the beginning, once again at the end of phase 1 (in the clinic) , and last time after home practice (the second phase).
DTVP-2 (developmental test of visual perception, 1993)) | Baseline
  Screening test.
Satisfaction questionnaire | up to 18 weeks